CLINICAL TRIAL: NCT00117416
Title: MAP and Renal Perfusion: Evaluation of Critically Ill Patients With Normal Creatinine or Reduced Renal Function
Brief Title: Mean Arterial Pressure (MAP) and Renal Perfusion: Evaluation of Critically Ill Patients With Normal Creatinine or Reduced Renal Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects recruited
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2002/382
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2021-07

CONDITIONS: Kidney Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: controlling the MAP

SUMMARY:
The purpose of this study is to evaluate the renal perfusion depending on the MAP.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Intensive care patient
* Treated with vasopressor
* Given informed consent
* Arterial infusion
* A bladder catheter

Exclusion Criteria:

* Anamneses of hypertension
* Neurological trauma
* Acute renal insufficiency other than prerenal or acute tubular necrosis etiology
* Hepatorenal syndrome
* Treated with diuretics
* Mechanical ventilation and unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-02; Primary Completion 2003-02; Study Completion 2003-02

PRIMARY OUTCOMES:
creatinine clearance after 4 hours

SECONDARY OUTCOMES:
resistance index
diuresis
urinary indices of renal function

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be